CLINICAL TRIAL: NCT03327662
Title: Utilising Circulating Tumour Cell (CTC) Counts to Optimize Systemic Therapy of Metastatic Prostate Cancer: CTC-STOP Trial
Brief Title: Utilising CTC Counts to Optimize Systemic Therapy of Metastatic Prostate Cancer
Acronym: CTC-STOP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Underrecruitment
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Prostate Cancer UK (Other); University of Twente (Other); Sanofi (Industry); Janssen, LP (Industry); Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2015/10054
Record Dates: First submitted 2017-10-10; First posted 2017-10-31 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Cabazitaxel; Docetaxel; Circulating Tumour Cells

STUDY DESIGN:
Intervention Model Description: Patients with CTC count >5 CTC/7.5 mL at screening will be randomised 1:1 to either the control group (standard of care) or intervention group (CTC guided treatment). All patients will commence first line chemotherapy with docetaxel 75mg/m2 three-weekly and will receive a minimum of 3 cycles of treatment before any recommendation to discontinue first-line docetaxel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Active CTC assessment: Patients will receive first line docetaxel until progression by CTC, and/or disease progression according to treating clinician or completion of 10 cycles. CTC results will be available to the treating clinician to guide decision-making. A progressing CTC count on Day 1 will require confirmation with a second CTC count performed on Day 15 (-/+ 5 days) of that cycle. If a patient is found to have two successive CTC determinations showing progression by CTCs, the clinician will receive a recommendation to discontinue docetaxel on the following cycle.
  Interventions: Other: Active CTC Assessment
- Control (No Intervention): Patients will receive first line docetaxel until disease progression according to treating clinician or completion of 10 cycles. Patients and treating clinicians will not be disclosed to the results of CTC determinations.

INTERVENTIONS:
Other: Active CTC Assessment — CTC Counts used to guide treatment switch
  Arms: Interventional

SUMMARY:
CTC-STOP is a multicentre prospective randomised controlled phase III trial for metastatic castration-resistant prostate cancer patients.

This study will determine if serial CTC counts can be used as early markers of progression to direct early discontinuation of docetaxel chemotherapy in patients with mCRPC without adversely impacting overall survival, when compared with standard approaches to guide treatment switch decisions.

DETAILED DESCRIPTION:
Patients with metastatic castration-resistant prostate cancer will be randomised 1:1 to either control group (standard of care) or intervention group (CTC-guided treatment). All patients will commence first line chemotherapy with docetaxel three-weekly and will receive a minimum of 3 cycles of treatment before any recommendation to discontinue first-line docetaxel.

* Control Group (standard of care): patients will receive first line docetaxel until disease progression according to treating clinician or completion of 10 cycles. Patients and treating clinicians will not be disclosed to the results of CTC determinations.
* Intervention Group (CTC guided treatment): patients will receive first line docetaxel until progression by CTC, and/or disease progression according to treating clinician or completion of 10 cycles. CTC results will be available to the treating clinician to guide decision-making. A progressing CTC count on Day 1 will require confirmation with a second CTC count performed on Day 15 (-/+ 5 days) of that cycle. If a patient is found to have two successive CTC determinations showing progression by CTCs, the clinician will receive a recommendation to discontinue docetaxel on the following cycle.

The reasons of the treating clinician to discontinue docetaxel will be reported in both groups. Patients who discontinue first line docetaxel according to the criteria for each group will be switched to second line chemotherapy with cabazitaxel. After progression on cabazitaxel or completion of 10 cycles, patients will be followed up for survival every three months until end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age ≥18 years
3. Histologically confirmed diagnosis of adenocarcinoma of the prostate with availability of archival tumour tissue for molecular analyses (small cell prostate cancer is an exclusion); if no histological diagnosis has ever been acquired a fresh bone marrow trephine tumour biopsy confirming the presence of CRPC must be pursued.

   o Tumour tissue blocks will be requested for processing. Sections will be cut with the blocks then returned to the referring hospital. If the block is not available, at least ten tumour tissue sections (formalin-fixed paraffin-embedded) at 5 microns each will be requested.
4. Metastatic castration-resistant disease with only bone metastases, confirmed by bone scan (within 4 weeks) or CT (within 6 weeks), of starting this trial (Cycle 1 Day 1). Patients with local recurrence, and bone metastases with an associated soft tissue component, will be allowed into the trial. Pelvic lymphadenopathy <1.5cm in short axis is not an exclusion.
5. Systemic chemotherapy indicated for disease progression, defined as:

   o Bone Scan Progression: Two or more new documented bone lesions over previous 6 months.

   AND/OR

   o Increasing serum PSA level: Two consecutive increases in PSA levels documented over a previous reference value obtained at least one week apart are required. If the third PSA value is less than the second, an additional fourth test to confirm the rising PSA is required.
6. Baseline laboratory values as stated below:

   * Creatinine ≤1.5 x upper limit of normal (ULN)
   * Bilirubin ≤1.0 x ULN
   * SGOT (AST) and SGPT (ALT) ≤2.5x ULN
   * Castrate serum testosterone level (<50 ng/dL-or-<1.7 nmol/L)
   * ANC ≥1.5 x 109cells/L
   * Platelet count ≥100 x 109/L
   * PSA ≥ 5ng/mL
7. CTC levels ≥ 5 cells / 7.5 mL
8. Prior treatment with abiraterone and/or enzalutamide, discontinued due to disease progression.
9. Patient willing to continue primary androgen suppression with gonadotropin-releasing hormone (GnRH) analogues (either agonists or antagonists) throughout the study, unless treated with bilateral orchiectomy.
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 (see Appendix A2).
11. At least 3 weeks should have elapsed since stopping any investigational agent at the time of randomisation. More than 4 weeks since completion of radiotherapy, other than when a single palliative fraction is administered when only a two week interval is required before trial treatment commencement.
12. Patient recovered from any therapy-related toxicity to ≤ grade 2, (except alopecia, anaemia and any signs or symptoms of androgen deprivation therapy).
13. Patient willing to comply with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
14. Participants must be surgically sterile or must agree to use effective contraception during the period of the therapy and for 12 months after the last dose of study treatment. Effective contraception is defined as double barrier contraception (e.g. condom plus spermicide in combination with a female condom, diaphragm, cervical cap or intrauterine device).

Exclusion Criteria

1. Received any prior cytotoxic chemotherapy as treatment for castration-resistant prostate cancer. Patients that have received chemotherapy for hormone-sensitive metastatic prostate cancer will be allowed onto the trial, if the patient merits retreatment with docetaxel and at least 12 months has elapsed since the patient has completed that previous docetaxel therapy.
2. Measurable soft tissue or lymph node metastases or any metastatic disease outside the bone that is RECIST measurable will be an exclusion (unless it is pelvic nodal disease <1.5cm in short axis). Bone metastases with associated soft tissue components will also not be an exclusion.
3. Received any cycling, intermittent or continuous hormonal treatment 28 days prior to randomisation with the exception of the continuous LHRH analogues.
4. History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated. Brain imaging for asymptomatic patients is not required.
5. Current symptomatic cord compression requiring surgery or radiation therapy. (Once the patient is successfully treated the patient will be considered eligible for the study).
6. Active second malignancy (except non-melanoma skin or superficial bladder cancer) defined as requiring anticancer therapy or within the previous two years.
7. Serious medical conditions such as heart failure, myocardial infarction, pulmonary thromboembolism within 12 months; stroke or treatment of a major active infection within 3 months of randomisation, as well as any significant medical illness that in the opinion of the Investigator would preclude protocol therapy.
8. Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device. Concomitant participation in observational studies is acceptable.
9. Hypersensitivity to the active substance, to any of its excipients (including polysorbate 80) or to other taxanes.
10. Concomitant vaccination with yellow fever vaccine
11. Concomitant use of medicinal products that are strong CYP3A inducers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  OS is defined as the time from the date of randomisation to the date of death (due to any cause). Patients alive at end of follow-up will be censored at the last documented date of follow-up.
  An initial non-inferiority analysis will be conducted followed by a superiority analysis if non-inferiority is demonstrated

SECONDARY OUTCOMES:
CTC-guided switch rates | 2 years
  Proportion of patients in the intervention group that undergo a chemotherapy switch from docetaxel to cabazitaxel guided by CTC results that fulfil the pre-specified criteria for progression.
CTC effects on chemotherapy | 2 years
  To determine if the study of serial CTC counts will decrease the administration of cytotoxic chemotherapy, number of cycles of chemotherapy in both groups will be reported.
Toxicity burden assessment | 2 years
  Incidence of treatment-emergent adverse events (safety and tolerability) will be assessed throughout the treatment period using the NCI CTCAE v4.0 and summarised in tabular format. Reported toxicities will be coded using MedDRA (current version)
Brief Pain Inventory | 2 years
  validated questionnaire that assesses pain severity (four items) and pain interference (11 items). Pain severity is measured through patients' rating of their level of current pain, average pain, least pain in the last 24 hours and worst pain in the last 24 hours, using an 11-point numerical rating scale (NRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The 'Worst Pain' and 'Average Pain' items of the BPI-SF are often used in clinical trials to singly represent pain severity.
The Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 2 years
  FACT-P is a relevant, worldwide Patient reported outcome measure tool used for assessing the health-related quality of life in men with prostate cancer. The FACT-P will be used in this study as part of a wider Quality of Life analysis to compare both arms.
EuroQoL Five Dimensions (EQ-5D) | 2 years
  EQ-5D is a self reported questionnaire measuring generic health status. EQ-5D will be used in this study as part of a wider Quality of Life analysis to compare both arms.
Progression Free Survival | 2 years
  PFS will be measured from the date of randomisation to the date of death (due to any cause) or disease progression (As per PCWG2 criteria), whichever occurs first. Patients alive and progression-free at the last documented date of follow-up will be censored at that date.
Radiographic Progression Free Survival (rPFS) | 2 years
  rPFS will be measured from randomisation to the occurrence of one of the following:
  1. Development of new nodal / soft tissue (inclusive of measurable soft tissue associated with lytic bone -metastases) lesions by CT as defined in RECIST 1.1 criteria, and/or
  2. Progression of bone disease by PCWG2 bone scan criteria and/or,
  3. Death of any cause
  In case of progression by bone scan, the date of progression will be considered as the date of the first bone scan showing new lesions.
Time to First Symptomatic Skeletal Related Event (SSRE) | 2 years
  The time to the first SSRE will be defined will be measured from the date of randomisation to the date of any of the following:
  1. First use of external-beam radiation therapy to relieve skeletal symptoms
  2. New symptomatic pathologic vertebral or non-vertebral bone fractures
  3. Spinal cord compression
  4. Tumour-related orthopaedic surgical intervention
  Patients alive and free of SSRE at the last documented date of follow-up will be censored at that date.
Time to CTC Progression | 2 years
  CTC progression will be based on serial CTC levels collected during the study. Time to CTC Progression will be defined as the time from randomisation to the time of first blood test showing progression by CTCs, defined by:
  1. Failure to achieve a 30% decline from Screening CTC counts (baseline) AND a failure to achieve a conversion from unfavourable (≥ 5 cells/7.5 mL) to favourable (< 5 cells/7.5 mL) count; or
  2. Conversion from favourable to unfavourable CTC counts after a previous CTC response; or
  3. A 30% increase in CTC count from nadir after a previous CTC response and an unfavourable CTC count (i.e. CTC ≥ 5 cells/7.5 mL).
  An additional CTC count will be required to confirm progression. If confirmed, the date of the first CTC count meeting criteria for progression will be used as progression date.
Circulating Tumour Cells (CTC) counts | 2 years
  Serial CTC levels collected during the study will be compared to evaluate the % CTC change from Screening (baseline). Change at any time point will be classified into response CTC (decline >30%), stable CTC (change between -30% and 30%) and progressive CTC (increase >30%).
  The endpoint of interest for this study is the proportion of patients with a stable CTC count by 12-weeks (or earlier if treatment discontinued).
Prostate Specific Antigen (PSA) Counts | 2 years
  PSA values will be measured at regular timepoints in the study. At each time point where PSA is measured, % change from baseline PSA value will be measured, maximum PSA decline at any time and decline after 12 weeks on 1st and 2nd line chemotherapy will be reported.
Rate of CTC Response | 2 years
  CTC response is defined by:
  1. A conversion from unfavourable (>= 5 CTC/7.5 mL) to favourable (< 5 CTC/7.5 mL) CTC counts OR
  2. A 30% or more decrease in CTC counts from screening (baseline).
Rate of Pain response | 2 years
  Pain response will be evaluated only in patients with a median BPI score of ≥2 and will be defined as a reduction of 2 points or more from baseline median BPI score without an increase in analgesic score maintained for 3 or more weeks.
  Pain Progression Pain progression will be defined as an increase of at least two-points in the worst pain score over the mean baseline score (as defined by the baseline BPI), maintained for at least two consecutive measurements approximately 3-weeks apart.
Health Economic assessment | 2 years
  A decision analytic model will be developed, modelling the CTC guided and comparator interventions. The model will analyse the most cost-effective strategy for the management of patients with progressive disease.

OTHER OUTCOMES:
Patient perception and preferences on therapeutic switch decisions. | 2 years
  Patient perception and preferences on therapeutic switch decisions will be assessed by the Treatment Switch Questionnaire, purposely designed by the study team.
Post-trial treatment options | 2 years
  Post-trial treatment will be collected for all patients during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, MBChB FRCP MSc PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (4):
- United Kingdom (4):
  - The Royal Marsden Hospital, Sutton, Surrey
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - University College London Hospital, London